CLINICAL TRIAL: NCT04238663
Title: A Randomised, Double Blind, Three-Arm, Single Dose, Parallel Study To Compare the Pharmacokinetics, Safety and Immunogenicity of MB02 (Bevacizumab Biosimilar Drug), US Licenced Avastin® and EU Approved Avastin® in Healthy Male Volunteers
Brief Title: Pharmacokinetic Study Comparing MB02 And US And EU Avastin® In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MB02 A 05 18
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MB02 (Bevacizumab Biosimilar) (Experimental): Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: MB02 (Bevacizumab Biosimilar)
- EU approved Avastin® (Active Comparator): Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: EU approved Avastin®
- US licenced Avastin® (Active Comparator): Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: US licenced Avastin®

INTERVENTIONS:
Drug: MB02 (Bevacizumab Biosimilar) — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90-minute infusion
  Arms: MB02 (Bevacizumab Biosimilar)
Drug: EU approved Avastin® — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90-minute infusion
  Arms: EU approved Avastin®
Drug: US licenced Avastin® — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90-minute infusion
  Arms: US licenced Avastin®

SUMMARY:
Randomized, double blind, parallel group, single dose, 3 arm study to investigate and compare the pharmacokinetics (PK), safety and immunogenicity profile of MB02 with US and EU Avastin® in healthy male subjects.

During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms. Safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

DETAILED DESCRIPTION:
The primary PK parameter endpoints are Cmax and AUC(0-∞) for bevacizumab. The secondary PK endpoints will include all other PK parameters for bevacizumab, including tmax, t1/2, CL and AUC(0-t).

The serum PK parameters of bevacizumab will be calculated using standard noncompartmental methods. An analysis of covariance model will be used to analyse the log-transformed primary PK parameters (AUC[0 ∞] and Cmax) and AUC(0-t). The model will include a fixed effect for treatment and body weight as a covariate.

All other PK parameters will not be subject to inferential statistical analysis.

Estimates of geometric mean ratios together with the corresponding 90% confidence intervals (CI) will be derived for the comparisons of the PK parameters as follows:

* MB02 versus EU Avastin®
* MB02 versus US Avastin®
* EU Avastin® versus US Avastin®

PK similarity will be achieved if the 90% CIs for the biosimilar-to-reference ratios of PK endpoints (AUC[0-∞] and Cmax) fall within the predefined 0.80-1.25 acceptance similarity criteria for all 3 pairwise comparisons; MB02 versus EU-approved Avastin®; MB02 versus US-licenced Avastin®; and EU-approved Avastin® versus US-licenced Avastin®.

All AEs will be listed and summarised using descriptive methodology. All observed, or patient-reported AEs will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The incidence of AEs for each treatment will be presented by severity and by association with the study drugs as determined by the Investigator (or designee). Each AE will be coded using the Medical Dictionary for Regulatory Activities. All safety data will be listed and summarised as appropriate.

Immunogenicity data (overall anti-drug antibody [ADA] incidence and titers, and neutralising ADA results) will be listed. A summary of the number and percent of subjects testing positive for ADA or neutralising antibodies (NAB) before the dose of MB02, EU Avastin®, or US Avastin® (Day -1) and at scheduled postdose assessments will be presented by treatment arm. All safety data and immunogenicity data summaries will be based on the safety analysis population. Select analyses may be repeated for subsets with or without ADA and de novo ADA formation as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Males of any race, between 18 and 55 years of age, inclusive, at Screening.
2. Body mass index between 18.5 and 29.9 kg/m2, inclusive, at Screening and Check-in.
3. Total body weight between 60 and 95 kg, inclusive, at Screening and Check-in.
4. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhaemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable) at Screening or Check-in as assessed by the Investigator (or designee).
5. Relevant clinical laboratory evaluations of haematology, coagulation, urinalysis and clinical chemistry within the following ranges at Screening and Check in. A single repeat test will be allowed at each timepoint.

   * Absolute neutrophil count ≥1.5 × 109 L
   * Platelet count ≥100 × 109 L
   * Haemoglobin >10 g/dl
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ ULN
   * Alkaline phosphatase (ALP) ≤1.5 × ULN
   * Total bilirubin ≤ 1.5 ULN with direct bilirubin <20% in case of total bilirubin > ULN
   * Blood urea nitrogen ≤1.5 × ULN
   * Creatinine <132.63 µmol/L
   * Serum albumin: ≥35 g/L
   * Total cholesterol ≤ 7.75 mmol/L
   * Triglycerides ≤ 3.42 mmol/L
   * Creatine kinase (CK) ≤3 × ULN
   * International normalised ratio (INR) 0.8 to 1.3
   * Urine dipstick for proteinuria <2+
6. Systolic blood pressure ≥90 mmHg and <140 mmHg and diastolic blood pressure ≥50 mmHg and <90 mmHg at Screening and Check in.
7. Subjects agree to use contraception.
8. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions. Subjects must have signed an informed consent before any study-related procedure or evaluation is performed.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. Any current or recent history of active infections, including localised infections. (Within 2 months prior Screening Visit for any serious infection which requires hospitalization or intravenous anti-infective, and within 14 days prior Screening Visit for any active infection which requires oral treatment).
4. History of, or planned surgery, including suturing, dental surgery or wound dehiscence within 30 days of dosing, or within 30 days of the last study visit.
5. Presence of a nonhealing wound or fracture.
6. Known history of clinically significant essential hypertension, orthostatic hypotension, fainting spells or blackouts for any reason, cardiac failure or history of thromboembolic conditions.
7. Medically significant dental disease or dental neglect, with signs and/or symptoms of local or systemic infection that would likely require a dental procedure during the course of the study.
8. Clinically relevant history of alcoholism, addiction or drug/chemical abuse prior to Check-in, and/or positive urinary test for alcohol or drugs of abuse at Screening or Check in.
9. History of bleeding disorders or protein C, protein S, and/or factor V Leiden deficiency.
10. History of clinically significant haemorrhage, epistaxis, GI bleeding, haemorrhoids and/or haemoptysis.
11. History of GI perforation, ulcers, gastro oesophageal reflux, inflammatory bowel disease, diverticular disease, or any fistulae.
12. Alcohol consumption of >24 units per week. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
13. Positive hepatitis panel, positive human immunodeficiency test. Subjects whose results are compatible with prior immunisation and not infection may be included at the discretion of the Investigator.
14. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to Check-in, or within 5 half lives of the investigational drug used in the study.
15. Use or intend to use slow-release medications/products considered to still be active within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
16. Use or intend use of any prescription medications/ nonprescription products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator or designee.
17. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
18. Have received a live or attenuated vaccine from 3 months prior to Screening or have the intention to receive a vaccine during the study.
19. Intend to travel to a region where a vaccination will be required due to endemic disease within 3 months of dosing.
20. Previous treatment with an anti VEGF antibody or any other protein or antibody targeting the VEGF receptor.
21. Use of tobacco- or nicotine-containing products within 1 year prior to Check-in, or positive cotinine test upon Screening or Check-in.
22. Receipt of blood products within 60 days prior to Check-in.
23. Donation of blood from 90 days prior to Screening, plasma from 14 days prior to Screening, or platelets from 42 days prior to Screening.
24. Poor peripheral venous access.
25. History of abnormal peripheral sensation including paraesthesia and/or numbness in arms and/or legs.
26. Have previously completed or withdrawn from this study or any other study investigating bevacizumab, and/or have previously received bevacizumab.
27. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.
28. Vulnerable subjects (e.g. persons kept in detention).
29. Subjects who are study site employees or immediate family members of a study site or Mabxience employee.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects may be enrolled
Enrollment: 115 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Sinn, MD, Principal Investigator — Early Phase Clinical Unit (EPCU) PAREXEL International GmbH
Locations (1):
- Early Phase Clinical Unit (EPCU) PAREXEL International GmbH, Berlin, Germany

REFERENCES:
- [Derived] Sinn A, Garcia-Alvarado F, Gonzalez V, Huerga C, Bullo F. A randomized, double blind, single dose, comparative study of the pharmacokinetics, safety and immunogenicity of MB02 (bevacizumab biosimilar) and reference bevacizumab in healthy male volunteers. Br J Clin Pharmacol. 2022 Mar;88(3):1063-1073. doi: 10.1111/bcp.15032. Epub 2021 Sep 4. PMID 34374114

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject in the US Avastin arm withdrew before receiving any study treatment.
Period: Overall Study
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Started | 38 | 38 | 38
Completed | 38 | 37 | 38
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin® | Total
Number analyzed (Participants) | 38 | 38 | 38 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (10.18) | 41.6 (11.10) | 38.3 (9.64) | 39.8 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 38 | 38 | 38 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 38 | 37 | 37 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 36 | 35 | 37 | 108
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.48 (2.723) | 24.59 (2.322) | 24.80 (2.712) | 24.62 (2.573)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Serum Concentration
Description: To compare the pharmacokinetic (PK) profiles of MB02, US Avastin® and EU Avastin® (in terms of Cmax) to establish bioequivalence between the 3 study arms. For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) for the geometric LS means ratios are fully contained within the predefined bioequivalence limits of 0.80 to 1.25.
Time Frame: Predose, 1.5 hours (end of infusion), 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 3-8, Day 10, Day 14, Day 21, Day 28, Day 42, Day 56, Day 78, and Day 100.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: (ng/mL)/(mg/mL)
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
(ng/mL)/(mg/mL) | 86100 (24.8) | 81100 (20.0) | 87500 (24.9)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (Cmax) falls completely within the range 0.80-1.25. The PK parameter Cmax was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of Geometric Least Square Mean = 1.06, 90% CI 2-sided [0.976 to 1.16] — For the comparison, MB02 represents the numerator and EU Avastin represents the denominator
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar) vs US Licenced Avastin®; For the comparison, MB02 represents the numerator and US Avastin represents the denominator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Mean = 0.983, 90% CI 2-sided [0.897 to 1.08]
Statistical Analysis 3: Comparison: EU Approved Avastin® vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Mean = 0.926, 90% CI 2-sided [0.851 to 1.01] — For Ratio of geometric least square mean (GLSM): EU is the numerator and US Avastin acts as the denominator

2. Primary Outcome: AUC(0-∞); Area Under the Serum Concentration-time Curve From Time Zero to Infinity
Description: To compare the pharmacokinetic (PK) profiles of MB02, US Avastin® and EU Avastin® (in terms of AUC[0-∞]) to establish bioequivalence between the 3 study arms. For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) for the geometric least square means (GLSM) ratios are fully contained within the predefined bioequivalence limits of 0.80 to 1.25.
Time Frame: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
ng*h/mL | 30700000 (16.2) | 28800000 (16.4) | 30700000 (12.9)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 0.80-1.25. The PK parameter AUC[0-∞] was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 1.07, 90% CI 2-sided [1.00 to 1.14] — For the comparison, MB02 represents the numerator and EU Avastin represents the denominator
Statistical Analysis 2: Comparison: MB02 (Bevacizumab Biosimilar) vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 0.998, 90% CI 2-sided [0.944 to 1.05] — For the comparison, MB02 represents the numerator and US Avastin represents the denominator
Statistical Analysis 3: Comparison: EU Approved Avastin® vs US Licenced Avastin®; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GLSM = 0.934, 90% CI 2-sided [0.884 to 0.988] — EU Avastin corresponds to the numerator and US Avastin corresponds to the denominator

3. Secondary Outcome: Tmax: Time of Maximum Observed Serum Concentration
Description: To evaluate and compare the tmax of MB02, US Avastin® and EU Avastin® .
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
hours | 4.0 [1.5 to 8.0] | 4.0 [1.5 to 11.9] | 4.0 [1.5 to 12.00]

4. Secondary Outcome: AUC(0 t)= Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Observable Concentration.
Description: To evaluate and compare the AUC[0-t] of MB02, US Avastin® and EU Avastin®.
Time Frame: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
ng*h/mL | 29900000 (15.6) | 27900000 (16.0) | 29900000 (12.5)

5. Secondary Outcome: CL: Total Body Drug Clearance After IV Administration
Description: To evaluate the CL of MB02, US Avastin® and EU Avastin®
Time Frame: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: l/hour
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
l/hour | 0.00770 (18.1) | 0.00823 (18.5) | 0.00766 (16.2)

6. Secondary Outcome: t1/2: Apparent Serum Terminal Elimination Half-life
Description: To evaluate the t1/2 of MB02, US Avastin® and EU Avastin®
Time Frame: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
hours | 443 (16.9) | 444 (14.5) | 458 (16.1)

7. Secondary Outcome: Immunogenicity: Number of Participants With Anti-bevacizumab Antibodies (Including Neutralizing Antibodies)
Description: Incidence of anti-bevacizumab antibodies (ADA), including neutralizing antibodies (Nab). Subjects who tested positive at baseline are not included here.
  Rows for ADA and nAb are not mutually exclusive, i.e. a participant could be included in more than one Row.
Time Frame: Day -1, Day 14, Day 28, Day 56, and Day 78
Measure: Number; unit: participants
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
participants
  ADA positive | 12 | 14 | 9
  NAb positive | 1 | 0 | 2

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (Safety)
Description: Compare the incidence of Treatment-emergent Adverse Events (TEAEs) reported in each treatment arm. TEAEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA version 22.0) and graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: Day 1 - Day 100
Measure: Number; unit: participants
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
participants
  Subjects with TEAEs | 30 | 25 | 32
  Subjects with SAEs | 0 | 0 | 0
  Subjects discontinued due to TEAEs | 0 | 0 | 0
  Not related TEAEs | 16 | 12 | 16
  Unlikely-related TEAEs | 4 | 2 | 4
  Possibly related TEAEs | 10 | 11 | 12
  TEAEs of mild severity | 20 | 10 | 23
  TEAEs of moderate severity | 10 | 14 | 9
  TEAEs of severe severity | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Study duration (Day 1 - Day 100)
Description: Coded according to Medical Dictionary for Regulatory Activities (version 22.0), and graded on the basis of the US National Cancer Institute's Common Terminology for Adverse Events (version 5.0).
  Following a request from the Medicines and Healthcare products Regulatory Authority (MHRA) all serious adverse reactions were considered unexpected and reported as SUSARs, for the purpose of safety reporting in healthy volunteers.
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | US Licenced Avastin®
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 30/38 | 25/38 | 32/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MB02 (Bevacizumab Biosimilar) (N=38) | EU Approved Avastin® (N=38) | US Licenced Avastin® (N=38)
Nasopharyngitis (Infections and infestations) | 14 (17) | 12 (12) | 13 (14)
Headache (Nervous system disorders) | 5 (6) | 9 (14) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (3) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Pulpitis dental (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04238663/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT04238663/SAP_003.pdf